CLINICAL TRIAL: NCT06715072
Title: Study on the Efficacy and Safety of Transarterial Chemoembolization Combined with Targeted Immunotherapy in Patients with Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Yao Xie (Other)
Responsible Party: Sponsor-Investigator, Yao Xie, professor, Beijing Ditan Hospital
Organization: Beijing Ditan Hospital (Other)
Other Study IDs: DTXY30
Record Dates: First submitted 2024-11-19; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Unresectable Liver Cancer
Keywords: Unresectable Liver Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a single-center, single-arm, prospective study. It enrolls patients with unresectable hepatocellular carcinoma (HCC). The study aims to investigate the efficacy and safety of transarterial chemoembolization combined with targeted immunotherapy in patients with unresectable HCC, providing treatment guidance for these patients.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) represents the sixth most common cancer and the third leading cause of cancer-related deaths worldwide. Hepatocellular carcinoma (HCC) accounts for 75% to 85% of PLC cases, with the main etiologies being hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Approximately 44-62% of HCC patients develop portal vein tumor thrombus (PVTT), which plays a major role in disease prognosis. These patients have a poor prognosis, with a median survival time of 2.7-4 months without any intervention, posing a significant challenge to clinicians. Both the National Comprehensive Cancer Network (NCCN) and the European Society for Medical Oncology (ESMO) guidelines recommend that HCC patients with PVTT be classified as Barcelona Clinic Liver Cancer stage C (BCLC-C) and receive systemic therapy.For unresectable HCC, trans-arterial chemoembolization (TACE) is one of the most commonly used techniques and can significantly improve survival rates. Compared to best supportive care, TACE can significantly extend the overall survival (OS) of PVTT type I-III HCC by nearly 3 months . Sorafenib, a tyrosine kinase inhibitor (TKI), is the first approved targeted drug and has shown some survival benefits in advanced HCC compared to placebo. The REFLECT trial demonstrated that lenvatinib improved time to progression (TTP) and objective response rate (ORR) compared to sorafenib [13]. Two other studies also confirmed that TACE combined with lenvatinib had significantly better clinical efficacy in HCC with PVTT compared to TACE combined with sorafenib.Increasing evidence suggests that immune checkpoint inhibitors (ICIs) combined with multi-kinase TKIs or vascular endothelial growth factor (VEGF) antibodies are becoming a trend in the treatment of advanced HCC. Moreover, the inflammatory factors produced and released during TACE treatment have a priming effect on adaptive immunity; TACE can induce spontaneous T-cell responses and modulate the tumor microenvironment. The combined use of TACE and ICIs may more effectively promote antitumor immune reconstitution. A retrospective study reported that TACE combined with camrelizumab and apatinib significantly improved OS in HCC, with an ORR superior to the dual regimen of apatinib and camrelizumab. Another retrospective study involving 22 patients with advanced HCC showed that using lenvatinib and camrelizumab with TACE could control tumor progression and extend survival. However, data on this triple regimen for treating unresectable hepatocellular carcinoma are limited. Therefore, this study will provide evidence for the triple regimen in treating unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:Voluntarily join this study and sign the informed consent form;Age ≥18 years and ≤68 years, receiving arterial chemoembolization combined with targeted immunotherapy, regardless of gender;At least one measurable lesion as defined by the Modified Response Evaluation Criteria in Solid Tumors (mRECIST);Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1;Child-Pugh score ≤7;Generally good condition, such as albumin >25 g/L, white blood cells >3×10^9/L (excluding causes such as hypersplenism), platelets >50×10^9/L, etc.;Expected survival >12 weeks;No fertility requirements.

Exclusion Criteria:Uncontrolled hypertension;Active autoimmune diseases;Concurrent other untreated malignancies;Pregnant or breastfeeding women;Active bleeding tendency or coagulation disorders;Severe liver, kidney, heart, or bone marrow dysfunction;Severe allergy to iodine contrast agents;Other contraindications to the use of TACE, lenvatinib, camrelizumab, atezolizumab, bevacizumab, etc.;The investigator believes that accompanying medical history may affect the subject's safe completion of the study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable Liver Cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Evaluation | tree years
  The time from the date of the first dose of lenvatinib to disease progression or death from any cause.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li M, Hao J, Jiang T, Deng W, Lu H, Wang S, Wan G, Xie Y, Yi W. Maternal and neonatal safety of COVID-19 vaccination during the peri-pregnancy period: A prospective study. J Med Virol. 2023 Jan;95(1):e28378. doi: 10.1002/jmv.28378. PMID 36478410